CLINICAL TRIAL: NCT04574388
Title: Evaluation of Open-Label Conditioned Placebo Analgesia for Postoperative Opioid Reduction Following Spinal Fusion
Acronym: COLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kristin Schreiber, Assistant Professor, Principle Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018P000854
Record Dates: First submitted 2018-12-06; First posted 2020-10-05 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Spine Surgery
Keywords: open label placebo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open label placebo (Active Comparator): participants will take open label placebo pills TID and in conjunction with other PRN analgesics
  Interventions: Other: open label placebo
- treatment as usual (No Intervention): participants will take PRN analgesics as usual

INTERVENTIONS:
Other: open label placebo — open label placebo pill
  Other Names: non-deceptive placebo
  Arms: open label placebo

SUMMARY:
This research aims to understand the impact of conditioned open label placebo (COLP) on opioid consumption and pain after surgery. The hypothesis being tested is that by pairing a non-deceptive placebo pill with regularly prescribed pain killers after surgery, will allow reduction in opioids taken while maintaining the same level of analgesia.

DETAILED DESCRIPTION:
Participants will be enrolled at preoperative clinic.

Inclusion criteria:

1. aged 18-75 years
2. scheduled for spinal fusion surgery
3. able to comprehend and willingness to participate in COLP
4. willingness to undergo psychophysical and psychosocial testing
5. willingness to participate in long-term follow-up.

Exclusion criteria:

1. delirium, psychosis, or other cognitive impairment limiting completion of study procedures
2. non-English speaking
3. contraindication to opioid usage

Preoperative psychosocial and pain questionnaires will be completed using a secure email link to REDcap, and brief quantitative sensory testing performed.

After completion of preoperative testing, they will be randomized to one of 2 treatments: COLP or treatment as usual (TAU).

Day of surgery: Patient will undergo scheduled spinal fusion and admitted for post-operative recovery as per normal surgical management. No restrictions on intraoperative anesthetics or post-operative pain management options will be made. Intraoperative medication use, including opioids, as well as post-operative opioid consumption and pain scores will be extracted from the medical record.

Inpatient and outpatient postoperative period: The study investigator or research assistant (RA) will train the participant and nursing staff in the self-administration of COLP with each analgesic administration in hospital, beginning on POD 0, pairing one open label placebo pill with each analgesic medication administration. Beginning on POD 2, patients will additionally be instructed to take a scheduled placebo pill at least 3 times/day, and in conjunction with their ongoing instances of PRN opioid utilization. Opioid administration and pain scores will be recorded in a daily diary, which the RA will help fill out on POD1 and 2 with them. At hospital discharge, the patients' bottle of placebo pills will be replenished. Patients will be instructed to continue scheduled and PRN use of opioids, and encouraged to use placebo pills. After discharge, the number of placebo and opioid pills that they use, as well as average pain at rest and with movement each day will be collected for up to 21 days via email linking to Redcap system. If preferred, patients will answer questions through daily SMS TEXT or telephone call, using a secure study phone. To protect patient's privacy there will be no identifiable information in the text messages. The SMS texts will be sent from a dedicated study phone that is MobileIron enabled. MobileIron is software used by Partners HealthCare that allows for more secure data management.

Follow-up visit: At surgical follow-up visit, patients will repeat baseline testing and participants in the COLP group will undergo a 15-minute semi-structured interview to determine the patient's experience with managing post-operative pain with COLP. Long term follow-up on pain, psychosocial impact and opioid use will be accomplished using the Redcap email survey system.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18-75 years, (2) scheduled for spinal fusion surgery up to, and including 4 levels, (3) able to comprehend and willingness to participate in COLP, (4) willingness to undergo psychophysical and psychosocial testing (5) willingness to participate in long-term follow-up.

Exclusion Criteria:

* (1) delirium, psychosis, or other cognitive impairment limiting completion of study procedures (2) non-English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
self administration of PRN opioids | day 3-17
  daily report of post-discharge opioid use in sub-acute postoperative period, converted into morphine milligram equivalents
acute postoperative pain | day 3-17
  daily brief pain inventory (BPI)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Schreiber, M.D., Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Flowers KM, Patton ME, Hruschak VJ, Fields KG, Schwartz E, Zeballos J, Kang JD, Edwards RR, Kaptchuk TJ, Schreiber KL. Conditioned open-label placebo for opioid reduction after spine surgery: a randomized controlled trial. Pain. 2021 Jun 1;162(6):1828-1839. doi: 10.1097/j.pain.0000000000002185. PMID 33449503